CLINICAL TRIAL: NCT02033993
Title: A Multicentre Randomized Phase II Trial Comparing Nab-Paclitaxel to Paclitaxel in Patients With Advanced Urothelial Cancer Progressing on or After a Platinum Containing Regimen.
Brief Title: Nab-Paclitaxel to Paclitaxel in Advanced Urothelial Cancer Progressing on or After Platinum Containing Regimen.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL12
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2020-10

CONDITIONS: Urothelial Cancer
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Nab-Paclitaxel - 260mg/m2: q21 days
  Interventions: Drug: Nab-Paclitaxel
- Arm 2 (Active Comparator): Paclitaxel - 175mg/m2: q21 days
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Nab-Paclitaxel
  Arms: Arm 1
Drug: Paclitaxel
  Arms: Arm 2

SUMMARY:
The purpose of this study is to compare the effects on urothelial cancer of nab-paclitaxel compared to paclitaxel to treat this disease.

This research is being done because currently there is no effective treatment for urothelial cancer that has progressed after prior chemotherapy.

DETAILED DESCRIPTION:
Nab-paclitaxel is a formulation of the chemotherapeutic drug paclitaxel that is combined with a human protein called albumin. In Canada, nab-paclitaxel is currently approved for the treatment of metastatic breast cancer. This drug has been tested in other cancers and has shown promising activity in lung cancer, melanoma and pancreatic cancer. Information from research studies suggests that nab-paclitaxel may be a useful treatment for urothelial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of TCC of the urinary tract (bladder, urethra, ureter, renal pelvis) and metastatic or locally advanced inoperable disease extent (T4, N2, N3 or M1 disease)

Note: Mixed histologies (except small cell) permitted if predominately TCC by IHC.

* Patients must have evidence of metastatic disease, but measurable disease is not mandatory. To be considered evaluable for the overall response rate (complete and partial response), patients must have at least one measurable lesion as follows:

  * X-ray, physical exam ≥ 20 mm
  * Conventional CT scan, MRI ≥ 20 mm
  * Spiral CT scan ≥ 10 mm
* Male or female, 18 years of age or older.
* ECOG performance status ≤ 2 at study entry
* Adequate hematological, renal and hepatic functions as defined by the following required laboratory values obtained within 14 days prior to randomization. If anemic, patients should be asymptomatic and should not be decompensated.

  * Absolute neutrophil count (ANC) ≥ 1.5 x10^9/L (1,500 cells/mm3)
  * Platelet count ≥ 90 x10^9/L (100,000/mm3)
  * Hemoglobin ≥ 90 g/L
  * Calculated creatinine clearance > 25 mL/min (Cockcroft and Gault formula)
  * Total bilirubin ≤ 1.5 times the upper limit of normal (≤ 2.5X if Gilbert's disease)
  * ALT (SGPT) ≤ 3 x ULN or ≤ 5 x ULN if hepatic metastases are present
* Patients may have had prior neoadjuvant or adjuvant therapy for completely resected disease, provided it was completed at least 12 months prior to randomization. Patients must have recovered from any acute toxic effects to ≤ Grade 2 from any prior treatments. Neoadjuvant or adjuvant chemotherapy will be considered to have been first line therapy in the metastatic setting if the patient progressed within 12 months of the last dose.
* Patients must have received one and only one prior chemotherapeutic regimen which included a platinum (at least one cycle) for metastatic/recurrent disease. Treatment must have been discontinued at least 4 weeks prior to randomization in this study. Patients must have recovered from any acute toxic effects to ≤ Grade 2 from any prior treatments
* Patients may not have had any prior therapy with a taxane in any setting.
* Patients may have had prior investigational agents but these must have been discontinued at least 4 weeks prior to randomization. Patients must have recovered from any acute toxic effects to ≤ Grade 2 from any prior treatments.
* Prior treatments with radiation therapy in the adjuvant and/or metastatic setting are permitted provided that at least 2 weeks have elapsed since the last fraction of radiation therapy and all treatment related adverse events are ≤ Grade 1 at the time of randomization.
* Patients may have had prior surgery provided that at least 4 weeks elapsed between the end of surgery and randomization onto the study. Patients must have recovered from any acute toxic effects to ≤ Grade 2 from any prior treatments.
* Patients may have peripheral neuropathy from previous treatments providing that it is ≤ Grade 1.
* Patient is able (i.e. sufficiently fluent) and willing to complete the health and demographic, quality of life, and health utilities questionnaires in either English or French. The baseline assessment must be completed within required timelines, prior to registration/randomization. Inability (illiteracy in English or French, loss of sight, or other equivalent reason) to complete the questionnaires will not make the patient ineligible for the study. However, ability but unwillingness to complete the questionnaires will make the patient ineligible.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days prior to randomization. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy, bilateral tubal ligation or vasectomy/vasectomized partner. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures.
* Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* In accordance with CCTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* A candidate for potentially curative surgery or radiotherapy.
* Patients with brain metastases are ineligible if they meet at least one of the following criteria:

  1. diagnosis within 3 months from randomization
  2. untreated brain metastases
  3. unstable brain metastasis as defined by:

     * cavitation or hemorrhage in the brain lesion
     * symptomatic state
     * daily prednisone or equivalent use greater than 10 mg

Patients do not need CT/MRI scans to rule out brain metastases unless there is a clinical suspicion of CNS metastases.

* Patients with serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:

  1. . any evidence of severe or uncontrolled systemic disease (i.e. known cases of hepatitis B or C or human immunodeficiency virus (HIV)).
  2. patients with active or uncontrolled infections.

     Screening for chronic conditions is not required, although patients known to have such conditions at screening should not be included.
* Women who are pregnant or breastfeeding.
* Patients with history of allergic or hypersensitivity reactions to any study drug or their excipients or with a history of allergic reactions attributed to compounds with similar chemical composition to any of the study drugs.
* Planned concomitant participation in another clinical trial of an experimental agent, vaccine or device. Concomitant participation in observational studies is acceptable.
* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years. Prior prostate cancer is allowed provided that it is an incidental finding at cystoprostatectomy with a PSA <0.5 ng/mL at randomization or a prior diagnosis of low risk prostate cancer at any time as defined by ≤T2, a Gleason Score of 6 or less and PSA <10 ng/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srikala Sridhar, Study Chair — Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario Canada
Locations (37):
- Australia (18):
  - Townsville Hospital, Douglas, Queensland
  - Nambour General Hospital, Nambour, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ashford Cancer Care Research, Kurralta Park, South Australia
  - Prince of Wales Hospital, Sydney, South Australia
  - Concord Cancer Centre, Sydney, South Australia
  - Liverpool Hospital, Sydney, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Peninsula Oncology Centre, Frankston, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Epworth Healthcare Freemasons Hospital, Richmond, Victoria
  - Western Hospital (renamed to Footscray Hospital), St Albans, Victoria
  - Border Medical Oncology (Murray Valley Private Hospital), Wodonga, Victoria
  - Royal Perth Hospital (renamed to Fiona Stanley Hospital), Perth, Western Australia
  - Port Macquarie Base Hospital, Port Macquarie
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - Hopital Charles LeMoyne, Greenfield Park, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sridhar SS, Blais N, Tran B, Reaume MN, North SA, Stockler MR, Chi KN, Fleshner NE, Liu G, Robinson JW, Mukherjee SD, Rahim Y, Winquist E, Booth CM, Nguyen NT, Beardsley EK, Alimohamed NS, McDonald GT, Ding K, Parulekar WR. Efficacy and Safety of nab-Paclitaxel vs Paclitaxel on Survival in Patients With Platinum-Refractory Metastatic Urothelial Cancer: The Canadian Cancer Trials Group BL.12 Randomized Clinical Trial. JAMA Oncol. 2020 Nov 1;6(11):1751-1758. doi: 10.1001/jamaoncol.2020.3927. PMID 32940628

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Nab-Paclitaxel - 260mg/m2: q21 days
  Nab-Paclitaxel
- Arm 2: Paclitaxel - 175mg/m2: q21 days
  Paclitaxel
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 99 | 100
Completed | 96 | 91
Not Completed | 3 | 9

BASELINE CHARACTERISTICS:
Population: ITT
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 99 | 100 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 43 | 81
  >=65 years | 61 | 57 | 118
Age, Continuous [Median (Full Range); unit: Years] | 67 [24 to 88] | 68 [35 to 84] | 67 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 70 | 74 | 144
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 79 | 81 | 160
  Australia | 20 | 19 | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: PFS is defined as the time from randomization to the first observation of disease progression or death due to any cause.
Time Frame: 42 months
Population: ITT population.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 99 | 100
Months | 3.35 [2.69 to 4.30] | 3.02 [2.14 to 4.40]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.31, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.92, 90% CI 2-sided [0.68 to 1.23]

2. Secondary Outcome: Overall Survival
Description: Time from randomization to the date of death due to any causes, or censored at last contact date.
Time Frame: 42 months
Population: ITT piopulation
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 99 | 100
Months | 7.46 [6.44 to 8.64] | 8.77 [6.11 to 10.61]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.40, Log Rank — 1-sided p-value; Hazard Ratio (HR) = 0.95, 90% CI 2-sided [0.70 to 1.30]

3. Secondary Outcome: Clinical Benefit Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started. Clinical Benefit Rate = OR + SD > 12 weeks.
Time Frame: 42 months
Population: ITT population
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 99 | 100
percentage of participants | 50.5 [42.2 to 58.8] | 43 [34.9 to 51.1]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.28, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.76 to 2.59]

4. Secondary Outcome: Time to Response
Description: Time from the date of randomkization to the date of objective response according to RECIST Response Criteria was first achieved.
Time Frame: 42 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 99 | 100
Months | 17.5 [5.49 to 17.5] | 35.8 [0.03 to 42]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p = 0.54, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.46 to 1.51]

5. Secondary Outcome: Health Related Quality of Life Evaluated Using EORTC-C15-Pal
Description: Quality of life will be assessed using the EORTC-C15-PAL questionnaire plus additional study specific questions.
  Changes in quality of life scores while on treatment (compared to baseline scores) will be examined using descriptive analyses and inferential statistics. The primary test to compare treatment arms will be the NCIC CTG Quality of Life Committee suggested response analyses. A change score of 10 points from baseline was defined as clinically relevant. Patients were considered improved if reported a score 10-points or better than baseline at any time point in QoL assessment. Conversely, patients were considered worsened if reported a score minus 10-points or worse than baseline at any time point in QOL assessment without the above-defined improvement being observed. Patients whose scores were between 10-point changes from baseline at every QoL assessment were considered as stable.
Time Frame: 42 months
Population: Patients with baseline and at least 1 after treatment evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 85 | 75
Participants
  Improved | 28 | 22
  Stable | 7 | 13
  Worsen | 50 | 40

ADVERSE EVENTS:
Time Frame: 42 months
Description: The CTC version 4.0
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 72/99 | 67/100
Serious Adverse Events (participants affected / at risk) | 28/99 | 19/100
Other Adverse Events (participants affected / at risk) | 96/99 | 97/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=99) | Arm 2 (N=100)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 1 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Fever (General disorders) | 0 | 3
Pain (General disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 1
Anaphylaxis (Immune system disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 4
Skin infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Other nervous system disorders (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 2
Other renal and urinary disorders (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=99) | Arm 2 (N=100)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 4
Hearing impaired (Ear and labyrinth disorders) | 3 | 8
Tinnitus (Ear and labyrinth disorders) | 5 | 5
Blurred vision (Eye disorders) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 19 | 29
Constipation (Gastrointestinal disorders) | 58 | 55
Diarrhea (Gastrointestinal disorders) | 34 | 27
Dyspepsia (Gastrointestinal disorders) | 10 | 9
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 8
Mucositis oral (Gastrointestinal disorders) | 14 | 8
Nausea (Gastrointestinal disorders) | 46 | 44
Vomiting (Gastrointestinal disorders) | 22 | 19
Chills (General disorders) | 7 | 2
Edema limbs (General disorders) | 22 | 22
Fatigue (General disorders) | 71 | 80
Fever (General disorders) | 15 | 13
Flu like symptoms (General disorders) | 10 | 3
Non-cardiac chest pain (General disorders) | 3 | 5
Pain (General disorders) | 9 | 12
Upper respiratory infection (Infections and infestations) | 4 | 9
Urinary tract infection (Infections and infestations) | 21 | 17
Weight loss (Investigations) | 14 | 9
Anorexia (Metabolism and nutrition disorders) | 46 | 44
Dehydration (Metabolism and nutrition disorders) | 9 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 34
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 16
Flank pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 9
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 12 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 22
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Other musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 29
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Dizziness (Nervous system disorders) | 16 | 6
Dysgeusia (Nervous system disorders) | 15 | 15
Headache (Nervous system disorders) | 13 | 13
Paresthesia (Nervous system disorders) | 10 | 3
Peripheral motor neuropathy (Nervous system disorders) | 6 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 72 | 64
Anxiety (Psychiatric disorders) | 17 | 17
Depression (Psychiatric disorders) | 7 | 12
Insomnia (Psychiatric disorders) | 37 | 24
Hematuria (Renal and urinary disorders) | 11 | 11
Other renal and urinary disorders (Renal and urinary disorders) | 1 | 5
Urinary frequency (Renal and urinary disorders) | 7 | 6
Urinary incontinence (Renal and urinary disorders) | 0 | 5
Urinary tract obstruction (Renal and urinary disorders) | 15 | 11
Urinary tract pain (Renal and urinary disorders) | 5 | 1
Pelvic pain (Reproductive system and breast disorders) | 12 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 27
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31 | 32
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 62 | 62
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 6
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 14
Hot flashes (Vascular disorders) | 5 | 6
Hypertension (Vascular disorders) | 6 | 3
Hypotension (Vascular disorders) | 5 | 1
Thromboembolic event (Vascular disorders) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-11-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT02033993/Prot_002.pdf
  • Statistical Analysis Plan (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02033993/SAP_000.pdf
  • Informed Consent Form (2014-12-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT02033993/ICF_001.pdf